CLINICAL TRIAL: NCT07122466
Title: Early Treatment ctDNA Dynamics to Predict Response to Chemotherapy in Patients With Advanced Pancreatic Cancer: a Prospective, Observational Pilot Study
Brief Title: Early Treatment ctDNA Dynamics to Predict Response to Chemotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0286
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tumor DNA circulating in the bloodstream (circulating tumor DNA; ctDNA) — ctDNA will be measured at the same times as CT scans (just before the start of treatment, as well as 2 months after), and the response measured by the ctDNA change will be compared to the response seen on the changes between the CT scans. The goal is to make sure that ctDNA response correlates well with CT scan response measurement.

SUMMARY:
This is a study that aims to understand whether a blood test measuring tumor DNA circulating in the bloodstream (circulating tumor DNA; ctDNA) shows a similar response as observed by a follow-up CT scan. To study this question, ctDNA will be measured at the same times as CT scans (just before the start of treatment, as well as 2 months after), and the response measured by the ctDNA change will be compared to the response seen on the changes between the CT scans. The goal is to make sure that ctDNA response correlates well with CT scan response measurement.

ELIGIBILITY:
Inclusion Criteria:

Prior/Concurrent Therapy Criteria

1. Patients must be initiating a new treatment regimen for pancreatic cancer at the time of their initiation in the study
2. Patients must have cytologic or histologic confirmation of pancreatic cancer
3. Patients must have measurable radiographic evidence of metastatic disease
4. Patients must be ≥18 years of age
5. Patients must have an ECOG Performance Status 0-2.
6. Patients must have adequate organ function for delivery of chemotherapy as evidenced by the following: Hgb ≥8 g/dL, platelets ≥ 75
7. Patients must not have renal dysfunction that would prevent administration of IV contrast for radiographic assessment.

   Regulatory Criteria
8. Patients must be informed of the investigational nature of this study and must sign and give written informed consent for this protocol in accordance with institutional and federal guidelines.
9. Patients of all races, genders, & ethnicities are eligible.

Exclusion Criteria:

No exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed sample size of 20 subjects is based on feasibility and availability of resources and not on a formal power calculation. The number of subjects is small, so as to quickly gather data that could inform a larger study.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
First follow-up imaging assessment | 2 months
  Compare first follow-up imaging assessment at 2 months with tumor response as assessed by ctDNA level change from baseline

SECONDARY OUTCOMES:
ctDNA Assessment Comparison | 2 months
  Compare ctDNA assessment at 2 months with earlier ctDNA measurements
Compare Signatera ctDNA test | 6 months
  Compare Signatera ctDNA test with another vendor
ctDNA, CA19-9, & CEA Response | 6 months
  Compare response of ctDNA with response of CA19-9 and CEA

OTHER OUTCOMES:
Exploratory - Organoid Samples | 2 months
  If organoid samples are available, compare drug response assessment from organoids to clinical response assessment at 2 months.
Exploratory - Sample Size | 6 months
  If sample size has enough power, to compare differences in early ctDNA response between regimens (FOLFIRINOX vs Gemcitabine-based treatment, at 3 days and 1 week, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel King, MD, Principal Investigator — Northwell Health
Locations (1):
- Zuckerberg Cancer Center, New Hyde Park, New York, United States